CLINICAL TRIAL: NCT07310108
Title: A Randomized Double-Blind Parallel-Group Placebo Controlled Clinical Trial of Cordyceps Militaris M2-116-04 for Its Potential Sport and Exercise Nutrition Applications in Healthy Active Adults
Brief Title: Evaluation of Cordyceps Militaris M2-116-04 for Its Potential Sport and Exercise Nutrition Applications in Healthy Active Adults
Acronym: FUN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB-25-28
Record Dates: First submitted 2025-12-04; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Aerobic; Exercise
Keywords: aerobic; exercise
MeSH Terms: conditions — Motor Activity | interventions — CMIP protein, Cordyceps militaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Placebo (maltodextrin) or Study Product (Cordyceps Militaris). The serving size is 3 capsules taken once per day, with or without food. The Placebo will match the Study Product in appearance, color, and format. All supplements will be in capsule form and provided by the sponsor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Product (Experimental): Cordyceps Militaris
  Interventions: Dietary Supplement: Cordyceps Militaris
- Placebo (Placebo Comparator): Placebo maltodextrin
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Cordyceps Militaris — Cordyceps Militaris Study Product
  Arms: Study Product
Other: Placebo — Maltodextrin placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effects of supplementation with Cordyceps militaris MS-116-04 on exercise performance, endurance, cardiovascular fitness, gastrointestinal wellness, mood, and recovery compared to a placebo in healthy active adults.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled trial will evaluate the effects of daily supplementation with Cordyceps militaris MS-116-04 on exercise performance, endurance, cardiovascular fitness, gastrointestinal wellness, mood, and post-exercise recovery in healthy, active adults.

Participants will complete five study visits over approximately four weeks. Before each visit, participants will follow standardized pre-visit controls, including an 8-10 hour fast, 12 hours without caffeine, nicotine, or alcohol, and 24 hours of no structured exercise.

Visit 1 (Screening/Familiarization) includes informed consent, medical and medication review, anthropometrics, body composition (InBody), screening questionnaires, and familiarization with all exercise testing procedures (VO2max/peak test, 30-minute cycling bout, and Time to Exhaustion [TTE] trial).

Visit 2 (Baseline Part A) includes medication review, questionnaires (SHS-GI, PANAS), adverse event monitoring, and a maximal cycling VO2max/peak test.

Visit 3 (Baseline Part B) includes resting blood samples (serum cortisol, amylase, TNF-α, IL-10), a 30-minute cycling bout at 60% VO2peak, a cycling TTE trial, Borg RPE, and additional blood sampling immediately and four hours post-exercise. A standardized carbohydrate snack is provided during the four-hour recovery period. Participants are then randomized and receive instructions for daily supplementation and compliance tracking.

Visit 4 (End-of-Study Part A; 28-30 days later) mirrors Visit 2 and includes questionnaires, adverse-event review, and a VO2max/peak test.

Visit 5 (End-of-Study Part B; ~72 hours later) replicates Visit 3, including all blood sampling, the 30-minute cycling bout, TTE trial, four-hour recovery period, and standardized snack. Supplement return and compliance calculations are completed at this visit.

ELIGIBILITY:
Inclusion Criteria:

Healthy males and females aged 20 to 50 years of age. Individual indicates they are currently engaged in and historically engaged in exercise (i.e., structured or unstructured) for the prior 12 months.

Subject has the ability to exercise on a cycle ergometer without issue or concern.

Subject has the ability to "sprint" (cycle Time to Exhaustion Trial) without any orthopedic or other limitations.

Body Mass Index (BMI) 19 to 29.9 kg/m2 (normal weight to overweight status) Subject is in good health and appropriate for exercise as determined by physical examination, medical history and the Physical Activity Readiness Questionnaire (PAR-Q).

Subject can exercise on a cycle ergometer without issue or concern. Subject is a non-smoker. Subject agrees to not use any new vitamin, mineral, or dietary supplement product until after study completion and to not take any vitamins, minerals or dietary supplements 24 hours prior to the exercise test visits.

Subject is willing and able to comply with the protocol including: attending the study scheduled appointments, of which two of the study visits may take up to five hours for completion.

Subject agrees to refrain from exercise for the 24 hours prior to any test visits.

Subject agrees to refrain from alcohol use for at least 24 hours before every study visit.

Subject agrees to refrain from using any antihistamines for the 24 hours prior to the exercise test visits.

Subject agrees to refrain from drinking any exercise recovery beverages during the study period.

Subject is able to understand and sign the informed consent to participate in the study.

Exclusion Criteria:

Subject has any of the following medical conditions: active heart disease, uncontrolled high blood pressure (≥ 140/90 mmHg), renal or hepatic impairment/disease, Type I or II diabetes, bipolar disorder, Parkinson's disease, unstable thyroid disease, immune disorder (such as HIV/AIDS), any medical condition deemed exclusionary by the Principal Investigator (PI) Subject has a history of cancer (except localized skin cancer without metastases) within 5 years prior to screening.

Subject has a medical condition or orthopedic problem making exercising on a cycle ergometer contraindicated.

Subject has a VO2 peak/max value above the following age/sex categorizations (as measured during Visit 1): Males 20-29y - 47.5 mL/kg/min, Males 30-39y - 46.0 mL/kg/min, Males 40-45y - 43.9 mL/kg/min, Females 20-29y - 41.0 mL/kg/min, Females 30-39y - 39.6 mL/kg/min, Females 40-45y - 38.1 mL/kg/min Subject is currently taking antihypertensives, hypoglycemic medications or stimulatory asthma medications.

Subject is on an unstable dose of medication (defined as fewer than 90 days at the same dose).

Subject is taking a prescription medication deemed exclusionary by the Principal Investigator (PI).

Subject has an allergy to any ingredients in the Study Product. Subject has a history of drug or alcohol abuse in the past 12 months. Subject has a history of a psychiatric illness requiring hospitalization in the past 12 months.

Subject has any condition or abnormality that in the expert opinion of the PI, participation in the study would compromise the safety of the subject or the quality of the study data.

Subject is participating in or has participated in another research study within 30 days prior to the Screening visit.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-05-21 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Change in Time to Exhaustion (TTE) | Baseline (Visit 3) to End of Study (Visit 5; approximately 4 weeks).
  To determine whether supplementation with Cordyceps militaris MS-116-04, compared to placebo, affects exercise performance as measured by change from baseline in cycling Time to Exhaustion (TTE), recorded in minutes and seconds.
Change in VO2max | Baseline (Visit 2) to End of Study (Visit 4; approximately 4 weeks).
  To determine whether Cordyceps militaris MS-116-04 affects cardiovascular fitness compared to placebo, as assessed by change in maximal or peak oxygen consumption (VO2max/peak) from baseline to the end of the study.
Change in Gastrointestinal Wellness (SHS-GI Score) | Baseline (Visit 2) to End of Study (Visit 4; approximately 4 weeks).
  To assess whether the Study Product, compared to placebo, impacts digestive and gastrointestinal wellness as measured by the change in Short Health Scale for Gastrointestinal Symptoms (SHS-GI) total score from baseline to end of study.
  The SHS-GI is a validated patient-reported outcome measure consisting of four items, each rated on a 7-point likert scale ranging from 1 to 7, resulting in a total score range of 4 to 28.
  * Higher scores indicate worse gastrointestinal symptoms and poorer gastrointestinal well-being.
  * Lower scores indicate fewer gastrointestinal symptoms and better gastrointestinal well-being.
Change in Mood States (PANAS Score) | Baseline (Visit 2) to End of Study (Visit 4; approximately 4 weeks)
  To evaluate whether Cordyceps militaris MS-116-04 influences mood compared to placebo, as assessed by change in Positive and Negative Affect Schedule (PANAS) scores.
  The PANAS is a validated self-report questionnaire consisting of 20 items, comprising two subscales: positive affect and negative affect. Each item is rated on a 5-point Likert scale ranging from 1 (very slightly or not at all) to 5 (extremely).
  * Positive affect subscale score range: 10 to 50. Higher scores indicate greater positive affect (better mood).
  * Negative affect subscale score range: 10 to 50. Higher scores indicate greater negative affect (worse mood).
Change in Stress Cortisol Across Recovery Period | Pre-exercise (resting), immediately post-exercise, and 4 hours post-exercise at baseline and after approximately 4 weeks of intervention.
  To determine whether the Study Product affects biomarker salivary cortisol measured at rest, immediately post-TTE, and four hours post-TTE.
Change in Salivary Amylase Across Recovery Period | Pre-exercise (resting), immediately post-exercise, and 4 hours post-exercise at baseline and after approximately 4 weeks of intervention.
  To determine whether the Study Product affects biomarker salivary amylase measured at rest, immediately post-TTE, and four hours post-TTE.
Change in TNF-α | Pre-exercise (resting), immediately post-exercise, and 4 hours post-exercise at baseline and after approximately 4 weeks of intervention.
  To determine whether the Study Product, compared to placebo, influences inflammatory responses as measured by salivary Tumor Necrosis Factor-alpha (TNF-α) collected pre-exercise, immediately post-exercise, and four hours post-exercise.
Change in IL-10 concentrations | Pre-exercise (resting), immediately post-exercise, and 4 hours post-exercise at baseline and after approximately 4 weeks of intervention.
  To determine whether the Study Product, compared to placebo, influences inflammatory responses as measured by Interleukin-10 (IL-10) collected pre-exercise, immediately post-exercise, and four hours post-exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Chad M Kerksick, PhD, Principal Investigator — Lindenwood University
Locations (1):
- Lindenwood University Exercise and Performance Nutrition Laboratory, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.